CLINICAL TRIAL: NCT03589885
Title: Multicenter, rAndomized, Double-blind, Placebo-conTrolled, 52-week stUdy to demonstRatE the Efficacy, Safety and Tolerability of Secukinumab Injections With 2 mL Auto-injectors (300 mg) in Adult Subjects With Plaque Psoriasis
Brief Title: Study of Efficacy and Safety of Secukinumab 2 mL Auto-injector (300 mg) in Subjects With Moderate to Severe Plaque Psoriasis
Acronym: MATURE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457A2325
Record Dates: First submitted 2018-07-05; First posted 2018-07-18 (Actual); Results first posted 2021-08-26 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Plaque Psoriasis
Keywords: Plaque psoriasis, auto-injector, 2 mL injection, secukinumab
MeSH Terms: interventions — secukinumab

STUDY DESIGN:
Intervention Model Description: A Phase IIIb 52-week multicenter, randomized, double-blind, placebo-controlled, parallel-group trial in approximately 120 subjects with moderate to severe plaque-type psoriasis
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Placebo 2 mL auto-injector (Placebo Comparator): Placebo to secukinumab s.c., provided in 2 mL auto-injector form
  Interventions: Drug: Placebo 2 mL auto-injector
- Placebo 1 mL prefilled syringe (Placebo Comparator): Placebo to secukinumab s.c., provided in 2 * 1 ml prefilled syringe form
  Interventions: Drug: Placebo 1 mL prefilled syringe
- Secukinumab 2 mL auto-injector (Experimental): Secukinumab 300 mg provided in 2 mL auto-injector form
  Interventions: Drug: Secukinumab 2 mL auto-injector
- Secukinumab 1 mL prefilled syringe (Active Comparator): Secukinumab 300 mg provided as 2x 1 mL prefilled syringe of 150 mg/mL
  Interventions: Drug: Secukinumab 1 mL prefilled syringe

INTERVENTIONS:
Drug: Placebo 2 mL auto-injector — All Placebo patients until week 8 (included): 2 mL auto-injector Placebo + 2x 1 mL prefilled syringe Placebo s.c. at randomization, weeks 1, 2, 3, 4 and 8.
  PASI 90 responders at week 12: 2 mL auto-injector placebo + 2x 1 mL prefilled syringe Placebo s.c. at weeks 12, 13, 14, 15, 16 and every 4 weeks thereafter until week 48.
  PASI 90 non-responders at week 12: 2 mL secukinumab 300 mg auto-injector + 2x 1 mL prefilled syringe Placebo s.c. at weeks 12, 13, 14, 15, 16 and 4-weekly thereafter until week 48
  Other Names: Placebo
  Arms: Placebo 2 mL auto-injector
Drug: Placebo 1 mL prefilled syringe — All Placebo patients until week 8 (included): 2 mL auto-injector Placebo + 2x 1 mL prefilled syringe Placebo s.c. at randomization, weeks 1, 2, 3, 4 and 8.
  PASI 90 responders at week 12: 2 mL auto-injector Placebo + 2x 1 mL prefilled syringe Placebo s.c. at weeks 12, 13, 14, 15, 16 and every 4 weeks thereafter until week 48.
  PASI 90 non-responders at week 12: 2x 1 mL secukinumab 150 mg prefilled syringe + 2 mL auto-injector Placebo s.c. at weeks 12, 13, 14, 15, 16 and 4-weekly thereafter until week 48
  Other Names: Placebo
  Arms: Placebo 1 mL prefilled syringe
Drug: Secukinumab 2 mL auto-injector — 2 mL secukinumab 300 mg auto-injector + 2x 1 mL prefilled syringe Placebo s.c. at randomization, weeks 1, 2, 3, 4, 8, 12, 13, 14, 15 , 16 and 4-weekly thereafter until week 48
  Arms: Secukinumab 2 mL auto-injector
Drug: Secukinumab 1 mL prefilled syringe — 2 x 1 mL secukinumab 150 mg prefilled syringe + 2 mL auto-injector Placebo s.c. at randomization, weeks 1, 2, 3, 4, 8, 12, 13, 14, 15, 16 and 4-weekly thereafter until week 48
  Arms: Secukinumab 1 mL prefilled syringe

SUMMARY:
The primary purpose of this study is to assess efficacy, safety and tolerability of a 2 mL pre-filled auto-injector (AI) of 300 mg secukinumab in patients with moderate to severe plaque psoriasis

DETAILED DESCRIPTION:
This is a 52-weeks multicenter, randomized, double-blind, placebo-controlled, parallel-group trial in approximately 120 subjects with moderate to severe plaque-type psoriasis

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for inclusion in this study must have fulfilled all of the following criteria:

1. Men or Women of at least 18 years of age at time of Screening
2. Subjects able to understand and communicate with the investigator and comply with the requirements of the study and must have given a written, signed and dated informed consent before any study related activity was performed. Where relevant, a legal representative signed the informed study consent according to local laws and regulations.
3. Chronic plaque-type psoriasis present for at least 6 months and diagnosed before Randomization.
4. Moderate to severe psoriasis as defined at Randomization by:

   * PASI score of 12 or greater, and
   * IGA mod 2011 score of 3 or greater (based on a scale of 0 - 4), and
   * Body Surface Area (BSA) affected by plaque-type psoriasis of 10% or greater.
5. Candidate for systemic therapy. This is defined as a subject having moderate to severe chronic plaque-type psoriasis that is inadequately controlled by

   * Topical treatment and/or
   * Phototherapy and/or
   * Previous systemic therapy

Exclusion Criteria:

1. Forms of psoriasis other than chronic plaque-type (e.g., pustular, erythrodermic and guttate psoriasis) at Screening or Randomization.
2. Ongoing use of prohibited treatments. Washout periods detailed in the protocol had to be adhered to. Subjects not willing to limit UV light exposure (e.g., sunbathing and/or the use of tanning devices) during the course of the study were considered not eligible for this study since UV light exposure was prohibited.

   Note: administration of live vaccines 6 weeks prior to Randomization or during the study period was also prohibited.
3. Previous exposure to secukinumab (AIN457) or any other biologic drug directly targeting IL-17 or the IL-17 receptor.
4. Use of other investigational drugs at the time of enrollment, or within 5 half-lives of enrollment, or within 30 days until the expected pharmacodynamic effect had returned to baseline, whichever is longer; or longer if required by local regulations.
5. Pregnant or nursing (lactating) women, where pregnancy was defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
6. History of lymphoproliferative disease or any known malignancy or history of malignancy of any organ system treated or untreated within the past 5 years, regardless of whether there was evidence of local recurrence or metastases (except for Bowen's disease, or basal cell carcinoma or actinic keratoses that had been treated with no evidence of recurrence in the past 12 weeks; carcinoma in situ of the cervix or non-invasive malignant colon polyps that have been removed).
7. History of hypersensitivity to any of study drug constituent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Actual)
Dates: Start 2018-12-19 (Actual); Primary Completion 2019-11-19 (Actual); Study Completion 2020-08-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (21):
- United States (8):
  - Novartis Investigative Site, Miami, Florida
  - Novartis Investigative Site, Marietta, Georgia
  - Novartis Investigative Site, Saint Joseph, Missouri
  - Novartis Investigative Site, Verona, New Jersey
  - Novartis Investigative Site, Portland, Oregon
  - Novartis Investigative Site, Houston, Texas
  - Novartis Investigative Site, San Antonio, Texas
  - Novartis Investigative Site, Sugar Land, Texas
- Canada (2):
  - Novartis Investigative Site, Edmonton, Alberta
  - Novartis Investigative Site, Surrey, British Columbia
- Germany (4):
  - Novartis Investigative Site, Bielefeld
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Vechta
  - Novartis Investigative Site, Witten
- Novartis Investigative Site, Kopavogur, Iceland
- Poland (2):
  - Novartis Investigative Site, Warsaw, Mazowian
  - Novartis Investigative Site, Wroclaw
- Spain (4):
  - Novartis Investigative Site, Alicante, Valencia
  - Novartis Investigative Site, Valencia, Valencia
  - Novartis Investigative Site, Barcelona
  - Novartis Investigative Site, Madrid

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- See also: A Plain Language Trial Summary is available on novartisclinicaltrials.com — https://www.novctrd.com/ctrdweb/patientsummary/patientsummaries?patientSummaryId=815

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 144 subjects were screened at 22 study centers in 6 countries, and 122 subjects were randomized.
Pre-assignment Details: A total of 144 subjects were screened at 22 study centers in 6 countries, and 122 subjects were randomized.
Groups:
- Secukinumab 300 mg (2 mL AI): Secukinumab 300 mg provided in 2 mL auto-injector form
- Secukinumab 300 mg (2x 1 mL PFS): Secukinumab 300 mg provided as 2x 1 mL prefilled syringe of 150 mg/mL
- Placebo: Placebo to Secukinumab
- Placebo-Secukinumab 300 mg (2 mL AI): Placebo patients up to Week 12 who thereafter received secukinumab in 2 mL AI up to the end of treatment
- Placebo-Secukinumab 300 mg (2 x 1 mL PFS): Placebo patients up to Week 12 who thereafter received secukinumab in 2 x 1 mL PFS up to the end of treatment
Period: Treatment Period 1-Randomized Set
Arm/Group | Secukinumab 300 mg (2 mL AI) | Secukinumab 300 mg (2x 1 mL PFS) | Placebo | Placebo-Secukinumab 300 mg (2 mL AI) | Placebo-Secukinumab 300 mg (2 x 1 mL PFS)
Started | 41 | 41 | 40 | 0 | 0
Completed | 41 | 39 | 37 | 0 | 0
Not Completed | 0 | 2 | 3 | 0 | 0
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Lack of Efficacy | 0 | 0 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 1 | 0 | 0
Period: Treatment Period 2-Randomized Set
Arm/Group | Secukinumab 300 mg (2 mL AI) | Secukinumab 300 mg (2x 1 mL PFS) | Placebo | Placebo-Secukinumab 300 mg (2 mL AI) | Placebo-Secukinumab 300 mg (2 x 1 mL PFS)
Started | 41 | 39 | 4 | 16 | 17
Completed | 40 | 34 | 3 | 16 | 16
Not Completed | 1 | 5 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 1 | 0 | 0 | 0
Not completed — Pregnancy | 1 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 3 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis set (FAS) consisted of 122 subjects and used for efficacy analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo | Total
Number analyzed (Participants) | 41 | 41 | 40 | 122
Age, Customized [Number; unit: Participants]
  < 65 | 39 | 37 | 36 | 112
  ≥ 65 | 2 | 4 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 12 | 37
  Male | 28 | 29 | 28 | 85
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 1
  Asian | 1 | 1 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 0 | 1
  White | 39 | 39 | 37 | 115
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: PASI 75 Response After 12 Weeks of Treatment
Description: Percentage of participants who achieve ≥ 75% reduction in PASI compared to baseline. A PASI (Psoriasis Area and Severity Index) score is a tool used to measure the severity and extent of psoriasis. The score ranges from 0 (no signs of psoriasis) to a theoretic maximum of 72. The intensity of redness, thickness and scaling of the psoriasis is assessed as none (0), mild (1), moderate (2), severe (3) or very severe (4).
Time Frame: 12 weeks
Population: Full Analysis Set: Set used for efficacy analysis (122 participants)
Measure: Number; unit: Participants
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo
Number analyzed (Participants) | 41 | 41 | 40
Participants | 39 | 34 | 4
Statistical Analysis 1: Comparison: Secukinumab 2 mL Auto-injector vs Placebo; PASI 75; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 1014.07, 95% CI 2-sided [68.83 to 14940.62]
Statistical Analysis 2: Comparison: Secukinumab 1 mL Prefilled Syringe vs Placebo; PASI 75; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 96.23, 95% CI 2-sided [17.22 to 537.78]

2. Primary Outcome: IGA Mod 2011 0 or 1 Response After 12 Weeks of Treatment
Description: Percentage of participants who achieve IGA mod 2011 0 or 1, and improved by at least 2 points on the IGA scale compared to baseline. This scale ranges from 0 (clear, no signs of psoriasis) to 4 (severe).
Time Frame: 12 weeks
Population: Full Analysis Set: Set used for efficacy analysis (122 participants)
Measure: Number; unit: Participants
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo
Number analyzed (Participants) | 41 | 41 | 40
Participants | 31 | 28 | 3
Statistical Analysis 1: Comparison: Secukinumab 2 mL Auto-injector vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 51.46, 95% CI 2-sided [11.95 to 221.64]
Statistical Analysis 2: Comparison: Secukinumab 1 mL Prefilled Syringe vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 29.70, 95% CI [7.38 to 119.57]

3. Secondary Outcome: PASI 90 Response
Description: Percentage of participants who achieve ≥ 90% reduction in PASI compared to baseline
Time Frame: 12 weeks
Population: Full Analysis Set: Set used for efficacy analysis (122 participants)
Measure: Number; unit: Participants
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo
Number analyzed (Participants) | 41 | 41 | 40
Participants | 31 | 26 | 2
Statistical Analysis 1: Comparison: Secukinumab 2 mL Auto-injector vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 88.46, 95% CI 2-sided [16.15 to 484.52]
Statistical Analysis 2: Comparison: Secukinumab 1 mL Prefilled Syringe vs Placebo; Test type: Superiority; p < 0.0001, Regression, Logistic; Odds Ratio (OR) = 37.90, 95% CI 2-sided [7.60 to 189.01]

4. Secondary Outcome: PASI 50, 75, 90 and 100 and IGA Mod 2011 0 or 1 Response
Description: Percentage of participants who achieve ≥ 50%, 75%, 90% and 100% reduction in PASI and achieve IGA mod 2011 0 or 1, and improved by at least 2 points on the IGA scale compared to baseline at each visit up to 52 weeks
Time Frame: 52 weeks
Population: Full Analysis Set: Set used for efficacy analysis
Measure: Number; unit: Participants
Groups:
- Placebo: Placebo to secuinumab
- Placebo-Secukinumab 300 mg (2 mL Auto-injector): Placebo patients up to Week 12 who thereafter received secukinumab in 2 mL aI up to the end of treatment
- Placebo-Secukinumab 300 mg (2x 1 mL Prefilled Syringe): Placebo patients up to Week 12 who thereafter received secukinumab in 2x 1mL PFS up to the end of treatment
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo | Placebo-Secukinumab 300 mg (2 mL Auto-injector) | Placebo-Secukinumab 300 mg (2x 1 mL Prefilled Syringe)
Number analyzed (Participants) | 41 | 41 | 40 | 16 | 17
Participants
  PASI 50 | 41 | 40 | 4 | 15 | 15
  PASI 75 | 38 | 37 | 1 | 13 | 14
  PASI 90 | 30 | 28 | 0 | 12 | 14
  PASI 100 | 23 | 18 | 0 | 11 | 11
  IGA 0/1 | 30 | 33 | 0 | 12 | 13

5. Secondary Outcome: Successful Self-injection
Description: Subject usability (ability to follow instructions for use and potential use-related hazards) and satisfaction with the new secukinumab 2 mL AI utilizing a self-administered Self-Injection Assessment Questionnaire (SIAQ) and investigator/site staff observation of secukinumab 300 mg 2 mL AI administration. The Satisfaction with Self-Injection (SA) domain score ranges from 0 (worst experience) to 10 (best experience).
Time Frame: From randomization until Week 28
Population: Safety Set was used for this analyses. For each visit only subjects with a value at both PRE-module at baseline and the respective POST-baseline visit are included.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- PRE- Module by Visit: PRE- Module by Visit score- Entire Treatment Period (Safety set)
- POST-module by Visit: POST-Module by Visit score-Entire Treatment Period (Safety Set)
- Absolute Change POST Module -PRE Module: Absolute Change POST Module -PRE Module scores
Arm/Group | PRE- Module by Visit | POST-module by Visit | Absolute Change POST Module -PRE Module
Number analyzed (Participants) | 122 | 122 | 122
Scores on a scale
  Baseline: number analyzed (Participants) | 114 | 0 | 0
  Baseline | 5.75 (2.442) |  |
  Baseline (1) =POST-module at baseline visit: number analyzed (Participants) | 113 | 113 | 113
  Baseline (1) =POST-module at baseline visit | 5.75 (2.452) | 7.52 (2.046) | 1.77 (2.789)
  Week 1: number analyzed (Participants) | 111 | 111 | 111
  Week 1 | 5.72 (2.463) | 8.11 (1.759) | 2.39 (3.169)
  Week 4: number analyzed (Participants) | 107 | 107 | 107
  Week 4 | 5.70 (2.495) | 8.27 (1.731) | 2.57 (3.080)
  Week 8: number analyzed (Participants) | 107 | 107 | 107
  Week 8 | 5.68 (2.490) | 8.62 (1.545) | 2.94 (2.869)
  Week 12: number analyzed (Participants) | 104 | 104 | 104
  Week 12 | 5.70 (2.523) | 8.56 (1.623) | 2.86 (2.985)
  Week 28: number analyzed (Participants) | 101 | 101 | 101
  Week 28 | 5.62 (2.485) | 8.69 (1.681) | 3.07 (3.238)

6. Secondary Outcome: Dermatology Life Quality Index, (DLQI) 0 or 1 Score (Total Score)
Description: DLQI is a simple, compact, and practical questionnaire for use in a dermatology clinical setting to assess limitations related to the impact of skin disease. The instrument contains ten items dealing with the participant's skin. With the exception of Item Number 7, the participant responds on a four-point scale, ranging from "Very Much" (score 3) to "Not at All" or "Not relevant" (score 0). Item Number 7 is a multi-part item, the first part of which ascertains whether the participant's skin prevented them from working or studying (Yes or No, scores 3 or 0 respectively), and if "No," then the participant is asked how much of a problem the skin has been at work or study over the past week, with response alternatives being "A lot," "A little," or "Not at all" (scores 2, 1, or 0 respectively). The DLQI total score is derived by summing all item scores, which has a possible range of 0 to 30, with 30 corresponding to the worst quality of life, and 0 corresponding to the best.
Time Frame: Change from Baseline up to 52 weeks
Population: Full Analysis Set-For each post-baseline visit only subjects with a value at both baseline and the respective post-baseline visit are included.
Measure: Mean (Standard Deviation); unit: Scores on a Scale
Arm/Group | Secukinumab 2 mL Auto-injector | Secukinumab 1 mL Prefilled Syringe | Placebo
Number analyzed (Participants) | 41 | 41 | 40
Scores on a Scale
  Week 12: number analyzed (Participants) | 38 | 40 | 37
  Week 12 | -13.21 (7.701) | -11.95 (7.861) | -1.97 (6.966)
  Week 28: number analyzed (Participants) | 41 | 40 | 3
  Week 28 | -13.59 (7.639) | -12.23 (8.438) | -13.00 (12.490)
  Week 52: number analyzed (Participants) | 41 | 40 | 3
  Week 52 | -12.44 (8.219) | -12.23 (8.408) | -14.33 (11.240)

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose of study treatment until end of study treatment (Week 48) plus 4 weeks post treatment.
Description: Any sign or symptom that occurs during the study treatment plus the 4 weeks post treatment.
Groups:
- Secukinumab 300 mg (2 mL Auto-Injector): Secukinumab 300 mg provided in 2 mL auto-injector form
- Secukinumab 300 mg (2 x 1 mL PFS): Secukinumab 300 mg provided as 2x 1 mL prefilled syringe of 150 mg/mL
- Any Secukinumab 300 mg (2 mL AI): Any Secukinumab 300 mg (2 mL AI)
- Any Secukinumab 300 mg (2 x 1 mL PFS): Any Secukinumab 300 mg (2 x 1 mL PFS)
- Placebo: Placebo to Secukinumab sub-cutaneous form
- Any Secukinumab 300 mg: Any Secukinumab 300 mg
Arm/Group | Secukinumab 300 mg (2 mL Auto-Injector) | Secukinumab 300 mg (2 x 1 mL PFS) | Any Secukinumab 300 mg (2 mL AI) | Any Secukinumab 300 mg (2 x 1 mL PFS) | Placebo | Any Secukinumab 300 mg
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/41 | 0/57 | 0/58 | 0/40 | 0/115
Serious Adverse Events (participants affected / at risk) | 1/41 | 3/41 | 1/57 | 4/58 | 0/40 | 5/115
Other Adverse Events (participants affected / at risk) | 19/41 | 16/41 | 24/57 | 21/58 | 5/40 | 45/115
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (2 mL Auto-Injector) (N=41) | Secukinumab 300 mg (2 x 1 mL PFS) (N=41) | Any Secukinumab 300 mg (2 mL AI) (N=57) | Any Secukinumab 300 mg (2 x 1 mL PFS) (N=58) | Placebo (N=40) | Any Secukinumab 300 mg (N=115)
Appendicitis (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 1 | 0 | 1 | 0 | 1
Device related infection (Infections and infestations) | 1 | 0 | 1 | 0 | 0 | 1
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0 | 1 | 0 | 1
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Secukinumab 300 mg (2 mL Auto-Injector) (N=41) | Secukinumab 300 mg (2 x 1 mL PFS) (N=41) | Any Secukinumab 300 mg (2 mL AI) (N=57) | Any Secukinumab 300 mg (2 x 1 mL PFS) (N=58) | Placebo (N=40) | Any Secukinumab 300 mg (N=115)
Nausea (Gastrointestinal disorders) | 0 | 3 | 0 | 3 | 0 | 3
Influenza like illness (General disorders) | 3 | 3 | 4 | 3 | 1 | 7
Nasopharyngitis (Infections and infestations) | 6 | 6 | 8 | 8 | 0 | 16
Upper respiratory tract infection (Infections and infestations) | 3 | 4 | 4 | 6 | 1 | 10
Headache (Nervous system disorders) | 2 | 4 | 3 | 4 | 1 | 7
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 2 | 3 | 3 | 2 | 6
Hypertension (Vascular disorders) | 4 | 2 | 5 | 2 | 0 | 7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-04-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT03589885/Prot_000.pdf
  • Statistical Analysis Plan (2018-11-23): https://cdn.clinicaltrials.gov/large-docs/85/NCT03589885/SAP_001.pdf